CLINICAL TRIAL: NCT02589405
Title: Benzaknen® 5% Gel in Combination With Dermotivin® Soft Liquid Soap and Non-comedogenic Cetaphil® Dermacontrol Moisturizer SPF30 in the Treatment of Mild-to-moderate Acne Vulgaris
Brief Title: Benzac 5% Gel in Combination With Cosmetic Products in Acne Vulgaris
Acronym: Benzac
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Collaborators: Proinnovera GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RD.03.SPR.105041
Record Dates: First submitted 2015-10-23; First posted 2015-10-28 (Estimated); Results first posted 2019-02-11 (Actual); Last update posted 2021-02-18 (Actual); Status verified 2018-09

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — Benzoyl Peroxide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Benzaknen treatment regimen (Experimental): Benzac® 5% Gel (once daily) + Dermotivin® Soft Liquid soap (twice daily) + Cetaphil® Dermacontrol Moisturizer SPF30 (once daily)
  Interventions: Drug: Benzoyl Peroxide; Other: Dermotivin® Soft Liquid cleanser; Other: Cetaphil® Dermacontrol Moisturizer SPF30

INTERVENTIONS:
Drug: Benzoyl Peroxide
Other: Dermotivin® Soft Liquid cleanser
Other: Cetaphil® Dermacontrol Moisturizer SPF30

SUMMARY:
The aim of this study is to evaluate a complete acne regimen consisting of a medication (Benzaknen® 5% Gel), and 2 cosmetic products Dermotivin® Soft Liquid soap and Cetaphil® Dermacontrol Moisturizer SPF30 in patients with acne.

DETAILED DESCRIPTION:
The main objective of this study is to evaluate subject satisfaction with the treatment regimen comprising Benzaknen® 5% Gel in association with 2 cosmetic products including a foam soap, Dermotivin® Soft Liquid soap, and a non comedogenic moisturizer, Cetaphil® Dermacontrol Moisturizer SPF30, in patients with mild to moderate acne, after 12 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subject of any ethnic background of 12 years or older.
* Subject with mild or moderate facial acne vulgaris defined as an Investigator Global Assessment (IGA) score at 2 or 3 on a 0-4 scale.
* Subject with any skin phototype according to T.B. Fitzpatrick skin phototype definitions.

Exclusion Criteria:

* Subject with severe acne (IGA>3) with nodules, cysts, scars or extra-facial lesions,
* Female subject who is pregnant, lactating or planning a pregnancy during the study,
* Subject susceptible to take a corticosteroid treatment during the study except inhaled or topic when needed to treat a condition outside the face,

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2015-08; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mi-Ran EGBERT, MD, Principal Investigator — Proinnovera GmbH
Locations (1):
- EGBERT Mi-Ran, Münster, Germany

REFERENCES:
- [Derived] Kim MR, Kerrouche N. Combination of benzoyl peroxide 5% gel with liquid cleanser and moisturizer SPF 30 in acne treatment results in high levels of subject satisfaction, good adherence and favorable tolerability. J Dermatolog Treat. 2018 Feb;29(1):49-54. doi: 10.1080/09546634.2017.1342758. Epub 2017 Jul 5. PMID 28678647

RESULTS

PARTICIPANT FLOW:
Groups:
- Three-part Treatment Regimen: Subject received a treatment regimen comprising Benzaknen® 5% Gel in association with Dermotivin® Soft Liquid cleanser and Cetaphil® Dermacontrol Moisturizer SPF30
Period: Overall Study
Arm/Group | Three-part Treatment Regimen
Started | 50
Completed | 46
Not Completed | 4
Not completed — Adverse Event | 3
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat population
Arm/Group | Three-part Treatment Regimen
Number analyzed (Participants) | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 21
  Between 18 and 65 years | 29
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 21.8 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33
  Male | 17
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Germany | 50
Skin phototype [Count of Participants; unit: Participants] — Skin phototype definitions according to T.B. Fitzpatrick. This was assessed by the investigator at baseline
  I: Always burns easily; never tans II: Always burns easily; tans minimally and with difficulty III:Burns minimally; tans gradually and uniformly (light brown) IV: Burns minimally; always tans well (moderate brown) V: Rarely burns; tans profusely (dark brown) VI: Never burns; deeply pigmented (black), tans profusely
  Participants
    Phototype I | 1
    Phototype II | 25
    Phototype III | 21
    Phototype IV | 3
Investigator Global Assessment [Count of Participants; unit: Participants] — IGA scale:
  0: Clear - Residual hyperpigmentation and erythema may be present
  1. Almost clear - A few scattered comedones and a few small papules
  2. Mild - Some comedones and some papules and pustules. No nodules present
  3. Moderate - Many comedones, papules and pustules.
  4. Severe - Covered with comedones, numerous papules and pustules and a few nodules may be present
  Participants
    Mild | 37
    Moderate | 13
    Severe | 0
Acne duration [Mean (Standard Deviation); unit: Years] | 9.8 (7.4)
Total lesion count [Mean (Standard Deviation); unit: Lesion] | 97 (45.6)
Non-Inflammatory lesions [Mean (Standard Deviation); unit: Lesions] — Definitions (assessment doned by trained investigator):
  Non-Inflammatory Lesions
  * Open Comedone: A mass of sebaceous material that is impacted behind an open follicular orifice (blackhead)
  * Closed Comedone: A mass of sebaceous material that is impacted behind a closed follicular orifice (whitehead)
  Inflammatory Lesions
  * Papules: A small, solid elevation less than one centimeter in diameter
  * Pustules: A small, circumscribed elevation of the skin which contains yellow-white exudate
  * Nodules/Cysts: A circumscribed, elevated, lesion generally more than 1.0 cm in diameter
  Lesions | 68.1 (37.2)
Inflammatory lesions [Mean (Standard Deviation); unit: Lesions] | 28.9 (21.7)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Satisfied and Very Satisfied With Regimen
Description: Number of subjects satisfied and very satisfied with the three-part treatment regimen
Time Frame: 12 weeks
Population: Only Data Observed: All subjects that answered this question (which explains the discrepancy with the total number of participants) -
Measure: Number; unit: participants
Groups:
- Treatment Regimen: Subjects treated with the three-part treatment regimen comprising Benzaknen® 5% Gel in association with Dermotivin® Soft Liquid cleanser and Cetaphil® Dermacontrol Moisturizer SPF30
Arm/Group | Treatment Regimen
Number analyzed (Participants) | 48
participants | 42

ADVERSE EVENTS:
Groups:
- Three-part Treatment Regimen: Subjects treated with the three-part treatment regimen comprising Benzaknen® 5% Gel in association with Dermotivin® Soft Liquid cleanser and Cetaphil® Dermacontrol Moisturizer SPF30
Arm/Group | Three-part Treatment Regimen
All-Cause Mortality (participants affected / at risk) | 0/50
Serious Adverse Events (participants affected / at risk) | 1/50
Other Adverse Events (participants affected / at risk) | 13/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Three-part Treatment Regimen (N=50)
Hypersensitivity (Immune system disorders) | 1 (1)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Three-part Treatment Regimen (N=50)
Laceration (Injury, poisoning and procedural complications) | 1 (1)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1)
Blepharitis (Immune system disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 (1)
Skin irritation (Skin and subcutaneous tissue disorders) | 3 (3)
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Herpes simplex (Infections and infestations) | 1 (1)
Impetigo (Infections and infestations) | 1 (1)
Mucosal infection (Infections and infestations) | 1 (1)
Nasopharyngitis (Infections and infestations) | 4 (4)
Pharyngitis (Infections and infestations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less